CLINICAL TRIAL: NCT03364673
Title: Stepping Into Survivorship: Harnessing Behavioral Economics to Improve Quality of Life in Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-361; CA166210 (Other Grant/Funding Number: NIH/NCI)
Record Dates: First submitted 2017-10-17; First posted 2017-12-06 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Physical Activity; Mobile Health; Fitness Tracker; Survivorship; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitness Tracker + Social Incentive Intervention (Experimental): Participants will enroll with a teammate (i.e. family or friend) and collaborate together. Teams will set a daily step goal, receive daily feedback on whether they achieved their goal, and receive a social incentive intervention.
  Interventions: Other: Fitness Tracker; Other: Social Incentive (Way to Health)

INTERVENTIONS:
Other: Fitness Tracker — Fitness trackers (e.g. Fitbit) are accelerometers that are worn on the wrist and tracks users' heart rate continuously in addition to steps, distance, calories, and active minutes
Other: Social Incentive (Way to Health) — The Way to Health platform is an automated information technology platform that integrates wireless devices, clinical trial randomization and enrollment processes, messaging (text, e-mail or voice), self-administered surveys, automatic transfers of financial incentives, and secure data capture for research purposes.

SUMMARY:
This research study will test whether using wearable fitness trackers with a social incentive, delivered through a game-based mobile health intervention, increases physical activity and quality of life in ovarian cancer survivors.

DETAILED DESCRIPTION:
Nearly 50% of ovarian cancer survivors experience poor quality of life, fatigue, and anxiety after completing surgery and chemotherapy to treat their disease. Moreover, many ovarian cancer survivors become deconditioned during treatment; 40% report significant drops in activity during the year after diagnosis, and only 20% meet the recommended guidelines for physical activity.

Interventional exercise studies are urgently needed to determine whether increasing physical activity improves outcomes in ovarian cancer survivors. In other cancers, physical activity improves quality of life and mental health, while reducing the risk of cancer recurrence and death. To date, however, most studies have focused on patients with curable breast and prostate cancers. The effects of physical activity on understudied populations, including ovarian cancer survivors, are unknown. Furthermore, although ovarian cancer survivors report an interest in participating in home-based walking programs, few formal programs exist.

Stepping into Survivorship is a single-arm study designed to test the effectiveness of a wearable fitness tracker with a game-based mobile health intervention that leverages social support to increase physical activity in ovarian cancer survivors. At the start of the study all participants will track their daily step counts using a wearable fitness tracker (e.g. Fitbit) to determine how many steps they walk in an average day. Next, they will set an increased step-goal and receive daily, individualized feedback based upon their performance.

Participants will also choose a team partner (i.e. family or friend) to receive a wearable fitness tracker and together they will track their steps, earning non-financial micro-incentives (e.g. points, levels, badges) when they achieve their collaborative goals. This game-based mobile health intervention is designed to enhance collaboration, accountability, peer support, and ultimately physical activity among ovarian cancer survivors and their friends/family members.

This research is being done to improve participants' quality of life. The investigators hope that the use of wearable fitness trackers with a game-based mobile health intervention will help participants increase their physical activity and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have newly diagnosed ovarian cancer
* Are ≤6 months of completing chemotherapy
* Read English
* Do not have cognitive, visual, or orthopedic impairments that would preclude participation
* Plan to continue treatment at Dana-Farber Cancer Institute

Exclusion Criteria:

* Participants will be excluded if they are already participating in an mHealth intervention
* Are unable to ambulate
* Do not have a smartphone to transmit data from the wearable tracker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A. Wright, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrier E, Xiong N, Thompson E, Poort H, Schumer S, Liu JF, Krasner C, Campos SM, Horowitz NS, Feltmate C, Konstantinopoulos PA, Dinardo MM, Tayob N, Matulonis UA, Patel M, Wright AA. Stepping into survivorship pilot study: Harnessing mobile health and principles of behavioral economics to increase physical activity in ovarian cancer survivors. Gynecol Oncol. 2021 May;161(2):581-586. doi: 10.1016/j.ygyno.2021.02.023. Epub 2021 Feb 23. PMID 33637350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fitness Tracker + Social Incentive Intervention
Started | 29
Completed | 24
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Injury unrelated to study | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 63 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Marital status [Count of Participants; unit: Participants]
  Married, partnered | 18
  Single | 4
  Widowed, separated | 2
International Federation of Gynecology and Obstetrics (FIGO) stage [Count of Participants; unit: Participants] — FIGO Stages range from I through IV. Median overall survival is greatest in early stage disease (IC and II) and worse is stage III-IV.
  Staging is determined using criteria such as the size of the tumor, if the cancer has spread to nearby lymph nodes, and if the cancer has spread to distant sites or organs.
  Participants
    IC | 5
    II | 1
    III | 1
    IIIB | 3
    IIIC | 6
    IVA | 3
    IVB | 5
Histology [Count of Participants; unit: Participants]
  Serous | 19
  Endometrioid | 3
  Carcinosarcoma | 1
  Clear cell | 1
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status
  0: Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  ECOG of 0 are considered to have fewer restrictions in their activities compared with those with an ECOG 1 or 2
  Participants
    0 | 5
    1 | 15
    2 | 4
Time from treatment completion to intervention enrollment, days [Mean (Standard Deviation); unit: days] | 45 (35)
Baseline daily steps [Mean (Standard Deviation); unit: steps] | 6210 (3328)
Teammate [Count of Participants; unit: Participants] — Self-selected family member or friend to participate as support partner
  Participants
    Spouse, partner | 11
    Sibling | 4
    Parent | 3
    Child | 2
    Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Accelerometer + Social Support + Gamification
Description: Feasibility will be defined as ≥60% of patients who participate in the pilot study complete the 24-week intervention
Time Frame: 1 year pilot
Population: Participants who initially consented to the study
Measure: Count of Participants; unit: Participants
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 29
Participants
  Completed intervention and follow-up period | 24
  Did not complete intervention and follow-up period | 5

2. Primary Outcome: Acceptability
Description: Study burden: To what extent do you agree or disagree with: "Participating in this study placed a substantial burden on me." (Options: strongly agree, agree, neutral, disagree, strongly disagree)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 24
Participants
  Participants indicate that the study was burdensome | 1
  Participants did not indicate that the study was burdensome | 23

3. Primary Outcome: Perceived Effectiveness
Description: To what extent do you agree or disagree with the following statements: "Participating in this study motivated me to increase my activity levels." Response options: strongly disagree, disagree, neutral, agree, strongly agree.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 24
Participants
  "strongly agree" or "agree" | 21
  "strongly disagree", "disagree", or "neutral" | 3

4. Secondary Outcome: Change in Daily Steps From Baseline to 12 Weeks
Description: To compare the change in daily steps from end of baseline to 12 weeks (after the end of baseline) to estimate outcome parameters for future study
Time Frame: 12 weeks [from end of baseline (day 15) to day 98]
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 24
steps
  Baseline (Day 1-14) | 6210.7 (3328.1)
  Intervention (Day 15-98) | 7643.0 (3610.9)

5. Secondary Outcome: Change in Daily Steps From Baseline 24 Weeks
Description: To compare the change in daily steps from end of baseline to 24 weeks (after the end of baseline) to estimate outcome parameters for future study
Time Frame: 24 weeks [from end to baseline (day 15) to day 182]
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Fitness Tracker + Social Incentive Intervention
Number analyzed (Participants) | 24
steps
  Baseline (Day 1-15) | 6210.7 (3328.1)
  Follow-up (Day 98-182) | 6435.1 (3550.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on an ongoing basis throughout the course of the study, Day 1-182.
Arm/Group | Fitness Tracker + Social Incentive Intervention
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
* Single-arm pilot study without a control group
* Participants were recruited from a single academic center, were required to have a smartphone, and needed to be able to identify a teammate. This may have resulted in the selection of a more affluent, educated, and socially-connected population than is representative of ovarian cancer survivors nationwide.
* We did not specifically measure other types of activity not captured by Fitbits (e.g., swimming or biking).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03364673/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03364673/ICF_001.pdf